CLINICAL TRIAL: NCT00115895
Title: Effect of the Radioiodine Dose in Thyroid Ablation- A Randomized Comparison of 1110 MBq to 3700 MBq
Brief Title: The Dose of Radioactive Iodine Needed to Ablate the Thyroid Remnant Left Behind After Thyroidectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Helsinki (Other)
Collaborators: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Hanna Mäenpää, Chief of Department, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYTJ001T/2000
Record Dates: First submitted 2005-06-26; First posted 2005-06-27 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: Thyroid Neoplasms
Keywords: radioiodine; serum thyroglobulin; whole body radioiodine scanning
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Iodine-131

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radioactive iodine 1,1 GBq (Experimental): Low activity of radioiodine, 1,1 GBq
  Interventions: Drug: Radioactive iodine
- Radioactive iodine 3,7 GBq (Other): Routine activity of radioiodine, 3,7 GBq
  Interventions: Drug: Radioactive iodine

INTERVENTIONS:
Drug: Radioactive iodine — Radioiodine is radionuclear treatment given in oral capsules in two activies 1,1 and 3,7 GBq
  Other Names: radioiodine

SUMMARY:
The thyroid cells take up iodine, and radioactive iodine is commonly used to irradiate residual thyroid tissue and thyroid cancer following surgical removal of the thyroid gland (thyroidectomy). A whole body radioactive iodine scanning is usually carried out after thyroidectomy to assess the amount of thyroid tissue left behind at surgery (that might still contain cancer), and to evaluate the presence of iodine avid lesions elsewhere in the body (that might be cancer metastases). A large dose of radioactive iodine is often given, still the optimal iodine dose to ablate the thyroid remnant after surgery is not known. In this study, two radioactive iodine doses are compared in the ablation of the thyroid remnant, a smaller (1110 MBq) dose and a larger (3700 MBq) dose. The study participants are randomly allocated using a 1:1 ratio to receive either the smaller or the larger radioactive iodine dose. These treatments are compared for safety, adverse effects, and the need for subsequent repeat treatments. The individual absorbed radiation doses are measured. The study hypothesis is that fewer repeat radioiodine treatments might be needed after the larger dose, but the larger dose might be associated with a higher frequency of adverse events.

DETAILED DESCRIPTION:
The study participants are randomly allocated to receive either a 1110 MBq or a 3700 MBq dose of radioiodine (131I) approximately 5 weeks after thyroidectomy. Thyroxin substitution is initiated only after administration of radioactive iodine. Treatment efficacy is monitored using serum thyroglobulin measurements and whole body radioiodine scanning. The absorbed radiation dose at the thyroid remnant and the biological half-life of radioactive iodine are measured with SPECT, 131I iodine detector and a Geiger counter.

Treatment related adverse events are collected using structured forms 4 to 5 days, 2 weeks and 3 months after administration of radioiodine. The need for a repeat treatment is assessed 4 to 6 months after the first administration of radioiodine. The criteria for a repeat radioiodine treatment are serum thyroglobulin > 1 ug/L and/or presence of abnormal radioiodine uptake in a whole body radioiodine scanning, which is carried out following a 4-week interruption of thyroxin supplementation or following administration of rhTSH.

Number of patients: 160

Aims of the study:

* To find out weather the risk for second radioiodine treatment differs with two dose levels of radioiodine: 1110 MBq or 3700 MBq.
* To study possible differences in the adverse effects in the treatment groups. Also days at hospital are counted.
* To analyse the effect of absorbed radiation dose to the treatment results

ELIGIBILITY:
Inclusion criteria:

* Total or near total thyroidectomy performed for papillary or follicular thyroid cancer
* R0-1 resection, no macroscopic cancer left behind at surgery
* Physically and emotionally able to undergo radioiodine treatment
* A written informed consent

Exclusion criteria:

* Pregnancy
* Physical or psychiatric illness that may deteriorate during the isolation period required by radioiodine therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2000-01; Primary Completion 2004-10 (Actual); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Cumulative number of radioactive iodine administrations | 15 yrs

SECONDARY OUTCOMES:
Adverse events | 15 yrs
Absorbed radiation dose | 15 yrs
Cancer recurrence | 15 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Hanna O Mäenpää, M.D. Ph.D., Principal Investigator — Deputy Chief Physician
Locations (1):
- Helsinki University Central Hospital, Department of Oncology, Helsinki, Finland

REFERENCES:
- [Background] Roos DE, Smith JG. Randomized trials on radioactive iodine ablation of thyroid remnants for thyroid carcinoma--a critique. Int J Radiat Oncol Biol Phys. 1999 Jun 1;44(3):493-5. PMID 10348276
- [Derived] Maenpaa HO, Heikkonen J, Vaalavirta L, Tenhunen M, Joensuu H. Low vs. high radioiodine activity to ablate the thyroid after thyroidectomy for cancer: a randomized study. PLoS One. 2008 Apr 2;3(4):e1885. doi: 10.1371/journal.pone.0001885. PMID 18382668
- See also: Helsinki University Central Hospital — http://www.hus.fi